CLINICAL TRIAL: NCT01716728
Title: Identification of Undiagnosed Lysosomal Acid Lipase Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Katherine Sims, MD, Neurologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012P000418
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Lysosomal Acid Lipase Deficiency; Cholesterol Ester Storage Disease
Keywords: Lysosomal Acid Lipase Deficiency; Cholesterol Ester Storage Disease; Wolman Disease; Lysosomal Storage Disorder; Metabolic Disease; Recessive Inheritance
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease; Lysosomal Storage Diseases; Metabolic Diseases | interventions — Restriction Mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzyme analysis (No Intervention): Patients invited for evaluation will undergo lysosomal acid lipase enzyme analysis
  Interventions: Other: enzyme analysis

INTERVENTIONS:
Other: enzyme analysis

SUMMARY:
Partners HealthCare maintains a Patient Data Registry (PDR) with information from all patient encounters at Partners HealthCare facilities. We intend to utilize the PDR to identify groups of patient who are of high clinical suspicion for undiagnosed lysosomal acid lipase deficiency. A group of potential participants will be identified through the PDR. Detailed records will be requested to further narrow to ideal participants based upon previously existing diagnoses and symptoms. Participants will be invited to partake in the study via a letter from their Partners care provider with supporting study details. Study participants will be evaluated in a one-time visit. A complete family and medical history will be collected. A physical exam will be performed, and up to 20cc of blood will be drawn. All participants will be notified of their disease status via letter and phone call from the study staff. If the study participant is diagnosed with LALD through this evaluation, proper follow-up recommendations and referrals will be provided. Our intent is to determine if existing patient data can successfully be utilized to aid in the identification of patients with rare genetic disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must have records available in the Partners HealthCare Patient Data Registry

Exclusion Criteria:

* Individuals must not have a diagnosis of Lysosomal Acid Lipase Deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
number of patients with previously undiagnosed GD identified Time Frame: up to 2 years Description: Safety Issue?: No number of patients with previously undiagnosed LALD identified | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Sims, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States